CLINICAL TRIAL: NCT07081854
Title: Effect of Aquatic Versus Land-Based Plyometric Exercises on Vertical Jump Performance and Landing Mechanics in Basketball Players
Brief Title: Aquatic Versus Land-Based Plyometric Exercises on Vertical Jump Performance and Landing Mechanics
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Sayed Abdelaziz Mohamed, principle investigator : mohamed sayed abdelaziz mohamed, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005756
Record Dates: First submitted 2025-07-02; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Healthy
Keywords: Basketball Players; Plyometric Exercises; Vertical Jump Performance; Landing Mechanics

STUDY DESIGN:
Intervention Model Description: Study group I and Study group II
Who Masked: Outcomes Assessor
Masking Description: sealed envelopes
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Land-Based Plyometric Training (Experimental): 20 Participants will perform traditional plyometric exercises on land (e.g., box jumps, depth jumps, jump squats)
  Interventions: Other: Land-Based Plyometric Training
- Aquatic Plyometric Training (Experimental): 20 Participants will perform plyometric exercises in a shallow pool (water depth ranging from the xiphoid process to just below it . The exercises will include water jump squats, water box jumps, and other water-resisted plyometric movements.
  Interventions: Other: Aquatic Plyometric Training
- General conditioning exercises (Active Comparator): 20 Participants will follow general conditioning exercises
  Interventions: Other: General conditioning exercises

INTERVENTIONS:
Other: Land-Based Plyometric Training — Participants will perform traditional plyometric exercises on land aimed at improving lower-body power and neuromuscular performance.
  Exercises:
  1. Box Jumps: Jumping onto a box of progressively higher levels to build explosive strength.
  2. Depth Jumps: Stepping off a box and immediately jumping vertically upon landing.
  3. Jump Squats: Explosive vertical jumps starting from a squat position.
  4. Lateral Bounding: Jumping side-to-side to enhance lateral agility.
  5. Broad Jumps: Maximal horizontal jumps for distance.
  6. Tuck Jumps: Jumping while bringing knees to the chest in mid-air.
  Arms: Land-Based Plyometric Training
Other: Aquatic Plyometric Training — Participants will perform plyometric exercises in a shallow pool, with the water depth fixed at the xiphoid process level (chest height). Greater peak mechanical power was observed for jumps performed in the water and was influenced by immersion depth.
  Exercises:
  1. Box Jumps: Jumping onto a box of progressively higher levels to build explosive strength.
  2. Depth Jumps: Stepping off a box and immediately jumping vertically upon landing.
  3. Jump Squats: Explosive vertical jumps starting from a squat position.
  4. Lateral Bounding: Jumping side-to-side to enhance lateral agility.
  5. Broad Jumps: Maximal horizontal jumps for distance.
  6. Tuck Jumps: Jumping while bringing knees to the chest in mid-air.
  Key Points:
  * Encouraged to perform movements explosively while applying maximal effort.
  * Proper execution is emphasized to maintain biomechanical integrity even in the water environment.
  * Water temperature: 25-28 °
  Arms: Aquatic Plyometric Training
Other: General conditioning exercises — Participants will follow a general conditioning routine that does not include plyometric exercises.
  Exercises:
  1. Bodyweight squats.
  2. Lunges.
  3. Core stability exercises (e.g., planks, bridges).
  4. General cardio activities such as light jogging or cycling.
  Arms: General conditioning exercises

SUMMARY:
This study will will be conducted to investigate the effect of aquatic versus land-based plyometric training on vertical jump performance, landing mechanics, quadriceps and hamstring muscles isometric strength in Basketball Players?

DETAILED DESCRIPTION:
Plyometric training, a type of exercise that involves explosive movements designed to enhance muscular power, has become a cornerstone in athletic conditioning. It is particularly effective for improving lower-body power and vertical jump performance, which are critical for sports such as basketball, volleyball, and track events. By utilizing the stretch-shortening cycle of muscles, plyometric exercises help athletes generate rapid force, thus enhancing their overall athletic performance. Vertical jump performance is a widely recognized indicator of an athlete's explosive power, agility, and lower-limb strength. In many sports, improving vertical jump height is prioritized as a key performance metric, as it reflects an athlete's ability to perform dynamic movements. Enhancements in jump height not only contribute to improved vertical leaps but also translate into better sprinting ability and more agile movements on the field.

While land-based plyometric training is well-established as an effective method for improving athletic performance, aquatic plyometric training has gained attention due to its low-impact nature. Although studies have compared these two modalities, there remains a lack of consensus regarding their relative effectiveness, necessitating further exploration Investigating how these different training methods influence athletic outcomes will help clarify their respective advantages and inform training practices. In contrast, aquatic plyometric training offers a lower-impact alternative by utilizing the buoyant properties of water. This training modality reduces the stress on joints and soft tissues while still enhancing jump performance. As a result, aquatic plyometric training is especially suitable for injury-prone athletes or those recovering from previous injuries, as the water's resistance can help improve strength without risking further harm.

While aquatic plyometric training may lead to smaller gains in vertical jump height compared to land-based training, it provides a safer environment for skill development. Studies have highlighted that aquatic training is especially beneficial for athletes who need joint protection, such as those involved in water sports. Its controlled environment helps mitigate the impact associated with high-intensity training, allowing athletes to maximize their performance without increasing injury risk. Proper landing mechanics are crucial to minimizing the risk of lower-extremity injuries during plyometric exercises. Faulty landing techniques, such as excessive knee valgus, are strongly linked to injuries like anterior cruciate ligament (ACL) tears. It is essential for training programs to incorporate biomechanical assessments to ensure that athletes execute movements safely, reducing the likelihood of injury.

Despite the valuable insights provided by recent research, further studies are needed to explore the effects of aquatic and land-based plyometric training across diverse athletic populations. Such research could inform the development of optimal training protocols that maximize performance and minimize injury risk.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 30 years old .
* Plyometric Training Experience: At least one year of prior experience in plyometric or athletic training.

Exclusion Criteria:

* Participation in any other exercise programs outside the experimental one (e.g., gymnastics).

  * History of severe musculoskeletal injuries or surgeries within the past 6 months.
  * Any medical conditions that would contraindicate plyometric exercise (e.g., cardiovascular, respiratory conditions).

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2026-05-10 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Vertical Jump height | up to 6 weeks
  Vertical jump height will be assessed using the My Jump smartphone application. This app utilizes the phone's camera and software to analyze jump height and velocity, providing additional data on jump performance.
vertival jumb velocity | up to 6 weeks
  Vertical jump velocity will be assessed using the My Jump smartphone application. This app utilizes the phone's camera and software to analyze jump height and velocity, providing additional data on jump performance.

SECONDARY OUTCOMES:
Landing Error Scoring System | up to 6 weeks
  Landing Error Scoring System is a clinical tool used to assess jump-landing mechanics for the video from my jumb land aplication . the feet, ankle, knees, hip, trunk, shoulder, neck and head posture is assessed through the video. it is a 17-item . According to the performance sheet, the questions 1-15 are Yes/No questions that are rated as 0 or 1. The questions 16 are rated as 0, 1, and 2; 0 = soft, 1= average and 2= stiff. the question 17 are rated as 0,1,2; 0= excellent,1 average and 2= poor, so the total score ranges from zero to 19. A higher score indicates poor technique in landing from a jump; a lower score indicates better jump-landing technique. the score are categorized as excellent which less than 4, good score more than four and less than or equal 5, moderate score less than four and poor more than six.
Quadriceps and hamstring strength | up to 6 weeks
  Quadriceps and hamstring strength will be measured using hand-held dynamometry. This portable device allows the examiner to assess isometric torque during maximal contractions of the muscles. It is effective for evaluating both proximal and distal muscles in all extremities. Studies consistently demonstrate high validity of hand held dynamometer measurements when compared to isokinetic dynamometers, especially for larger muscle groups such as the quadriceps and hamstrings. It was found that hand held dynamometer correlates strongly with isokinetic dynamometry (correlation coefficients r = 0.84-0.97) for measuring quadriceps and hamstring strength.